CLINICAL TRIAL: NCT03881241
Title: Multicenter, Post-market Observational Study Evaluating Safety and Efficacy of the EVOS SMALL Plating System for the Treatment of Lower Extremity Fractures
Brief Title: Safety Study of Treatment of Leg Fractures
Acronym: EVOS SMALL
Status: Terminated | Type: Observational
Why Stopped: Difficulty with enrollment
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018.18.TMA.EVOSM.PRO.EXT
Record Dates: First submitted 2019-03-11; First posted 2019-03-19 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Tibial Fractures
Keywords: Tibia; fracture; EVOS; EVOS SMALL; plating system; plates; tibial fracture; surgery; open reduction; internal fixation
MeSH Terms: conditions — Tibial Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Study Treatment: EVOS SMALL PLating System

SUMMARY:
This study evaluates the safety of the EVOS SMALL Plating system in patients who have a fracture of the tibia requiring surgery.

DETAILED DESCRIPTION:
This is a multicenter, prospective, post-marketing, observational, case series study to evaluate the safety and efficacy of the EVOS SMALL Plating System in subjects with proximal or distal (pilon or ankle) tibial fractures. Subjects will be recruited in the hospital emergency room or surgical department, at the point of identification of the need for ORIF surgery, and the decision is made to use the EVOS SMALL Plating System. The choice of medical and surgical treatment will be made independently by the Investigator in the regular course of practice and will not be influenced by this study protocol.

Approximately 100 subjects will be enrolled in order to ensure at least 90 evaluable subjects, with a minimum of 45 evaluable subjects having either a) proximal or b) distal tibial fractures.

Safety monitoring will include documentation device- and surgery-related AEs. Efficacy will be monitored by assessment of post-operative fracture resolution according to standard radiological practice (X-rays), clinical complications, reoperation rate, DRI, EQ-5D-5L, and pain VAS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject who is 18 years of age or older at the time of signing the informed consent.
2. Subject provides an Institutional Review Board (IRB)-approved informed consent. The subject must have the physical and mental capacity to provide informed consent for him/herself.
3. Subject has experienced proximal tibial fracture (OTA Type 41 A-C) or distal tibial fracture (OTA 43 Type A-C) with or without fibular/malleolar involvement (OTA 44 A-C) and are scheduled for ORIF using the EVOS SMALL Plating System.
4. Subject is willing and able to attend all study visits including 1 year post-operative follow-up.

Exclusion Criteria:

1. Subject has contraindications or hypersensitivity to the use of the EVOS SMALL Plating System or its components (316L stainless steel).
2. Subject has a physical condition that, in the opinion of the Investigator, would preclude adequate implant support or retard healing, such as blood supply impairment, insufficient bone quality or quantity, previous infection, obesity, severe bow or gross bony distortion of the tibia, as detailed in the IFU.
3. Subject has, in the opinion of the Investigator, an emotional or neurologic condition that precludes cooperation and compliance with the rehabilitation regimen.
4. Subject is currently in another investigational drug, biologic, or device study or has been treated with an investigational product within the last 30 days.
5. Subject is known to be at risk for loss to follow-up, or failure to return for scheduled visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years and older having either proximal or distal tibial fractures.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Reoperation rate for any reason of the lower extremity fractures treated operatively with the EVOS SMALL Plating System | 1 year

SECONDARY OUTCOMES:
Number of adverse events | 1 year
Disability Rating Index (DRI) | 1 year
  Change in subject's ease of mobility as marked on a 100 mm line by subject with the far left indicating "without difficulty" and the far right indicating "not at all"
EuroQoL-5D Questionnaire | 1 year
  Change in quality of life from baseline to one year postoperatively by answering quality of life questions on a 1-5 scale with 1 representing "never" and 5 representing "always"
Pain using visual analog scale (VAS) | 1 year
  level of pain as marked on a 100 mm line by subject with 0mm representing "no pain" and 100mm representing "worst possible pain"
Number of complications relating to surgery | 1 year
Number of hospital readmissions for any reason | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Nelson, Study Chair — Smith & Nephew, Inc.
Locations (2):
- United States (2):
  - Athens Orthopedic Clinic, Athens, Georgia
  - John Peter Smith Hospital, Fort Worth, Texas